CLINICAL TRIAL: NCT01800864
Title: Leptin Biology in Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, PI, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11-003834
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal (Other): Normal weight subjects
  Interventions: Other: obesity
- Over weight /obese subjects (Other): Overweight and obese subjects
  Interventions: Other: obesity

INTERVENTIONS:
Other: obesity

SUMMARY:
Leptin is a fat hormone which acts in maintaining energy balance. However, leptin levels are high in obese subjects indicating resistance to the actions of leptin. High leptin levels have been associated with increased cardiovascular and metabolic risks, but it is not clear if increased leptin or leptin resistance contributes to the increased cardiovascular risk. Further, even though leptin receptors are present in fat tissue, leptin's role in fat tissue functions are not completely investigated in humans. Based on preliminary data the investigators hypothesize that resistance to leptin action in obese adipose tissue is responsible for altering the expression of adipose tissue proteins which contribute to the development of cardiovascular and metabolic dysfunction. To test this hypothesis the investigators propose a novel study directed at investigating the leptin dependent changes in adipose tissue protein expression using adipose tissue obtained from lean and obese human subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. BMI BMI ≤25 (lean) or >30 kg/m2 (obese)
3. Going to undergo a surgical procedure where omental and subcutaneous adipose tissue may be biopsied.

Exclusion Criteria:

Inability to provide written informed consent.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Changes in adipose tissue protein expression in response to leptin treatment | Baseline and after 24 hours of leptin treatment
  The effect of leptin on adipose tissue protein expression will be assessed by Western blot method. The adipose tissue biopsy samples will be treated with leptin for 24 hours in sterile culture conditions. After leptin treatment, the tissue will be lysed, proteins will be separated by denatured SDS-PAGE electrophoresis, transferred on a nitrocellulose membrane and changes in specific proteins will be determined using protein-specific antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Virend K Somers, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States